CLINICAL TRIAL: NCT01298102
Title: Safety and Efficacy of Influenza A/H1N1/2009-adjuvanted Vaccine in Renal Transplant and Dialyzed Patients: a Prospective Cohort Study.
Brief Title: Influenza A/H1N1/2009-adjuvanted Vaccine in Renal Disease Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Broeders Nilufer, Hospital Erasme
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Etude 2009/INT044
Record Dates: First submitted 2011-02-16; First posted 2011-02-17 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2010-06

CONDITIONS: Decreased Immunologic Activity [PE]; Influenza; Rejection
Keywords: kidney; transplantation; haemodialysis; vaccination; influenza H1N1 2009
MeSH Terms: conditions — Influenza, Human; Rejection, Psychology | interventions — pandemrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- influenza vaccine (Experimental): Pandemrix vaccine (Influenza A/H1N1 2009)to be injected to renal transplant patients, haemodialyzed patients, and controls
  Interventions: Biological: Influenza A/H1N1 2009-AS03 adjuvanted (Pandemrix)

INTERVENTIONS:
Biological: Influenza A/H1N1 2009-AS03 adjuvanted (Pandemrix) — intramuscular injection of 1 dose vaccine
  Other Names: Pandemrix

SUMMARY:
In 2009, the pandemic influenza A/H1N1 accounted for worldwide recommendations about vaccination. There is no data concerning the immunogenicity nor the security of the adjuvanted-A/H1N1 vaccine in renal disease patients. The aim of this study is to observe the effects of this vaccine on transplanted and hemodialyzed patients.

DETAILED DESCRIPTION:
The serologic responses to the Pandemrix vaccine will assess the efficacy, with the determination of the seroconversion rate among the patients.

The anti-HLA and anti-MICA antibodies will be determined to assess the safety among the renal transplanted patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients
2. Haemodialyzed patients
3. Renal transplant recipients who have stable renal function for the last 3 months

Exclusion Criteria:

1. No pneumonia or severe infection during 1 month before vaccination
2. No Ivig (intravenous immunoglobulins) treatment during the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
to determine the efficacy aand safety of influenza A/H1N1 adjuvanted-vaccination among renal transplant and haemodialyzed patients as compared to controls | one month post-vaccination
  measures of anti-A/H1N1 antibodies with a method of microneutralizing test (seroneutralization) to follow-up the secondary effects of the vaccine and follow-up of renal function in renal transplanted patients.

SECONDARY OUTCOMES:
to controls and to assess the safety of the vaccine among renal transplanted patients by studying HLA or MICA sensitization before and following vaccination | follow-up 6 months
  To measure the Anti-HLA and anti-MICA antibodies with luminex-test

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Abramowicz, PhD, Study Director — Hospital Erasme
Locations (1):
- Hospital Erasme, Brussels, Brabant, Belgium

REFERENCES:
- [Background] Candon S, Thervet E, Lebon P, Suberbielle C, Zuber J, Lima C, Charron D, Legendre C, Chatenoud L. Humoral and cellular immune responses after influenza vaccination in kidney transplant recipients. Am J Transplant. 2009 Oct;9(10):2346-54. doi: 10.1111/j.1600-6143.2009.02787.x. Epub 2009 Jul 28. PMID 19656126